CLINICAL TRIAL: NCT06589271
Title: A Clinical Research on SCLife®-LDD hUC-MSCs Injection Therapy for Patients With Lumbar Intervertebral Disc Degeneration
Brief Title: SCLife®-LDD hUC-MSCs Injection Therapy for Patients With Lumbar Intervertebral Disc Degeneration
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of financial support
Sponsor: Sclnow Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCLnow-SH-01
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Lumbar Disc Degeneration
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Intervention Model Description: non-randomized, self-controlled, single-dose
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hUC-MSCs transplantation group (Experimental): Human Umbilical Cord Mesenchymal Stem Cells
  Interventions: Biological: human umbilical cord mesenchymal stem cell suspension
- control group (Active Comparator): suspension transplantation
  Interventions: Procedure: total endoscopic extraction of lumbar nucleus pulposus

INTERVENTIONS:
Biological: human umbilical cord mesenchymal stem cell suspension — 2 * 10^7 cells (2ml)
  Arms: hUC-MSCs transplantation group
Procedure: total endoscopic extraction of lumbar nucleus pulposus — hUC-MSCs are injected into the opposite side of the minimally invasive surgical site immediately after surgery, and the puncture needle remains for 1 minute after injection and then pull out to prevent cell suspension leakage
  Arms: control group

SUMMARY:
In recent years, total endoscopic extraction of nucleus pulposus has been widely used in the treatment of lumbar disc herniation due to its advantages of less trauma, faster recovery and less cost. However, the residual nucleus pulposus may protrude again after extraction, and the stability of the operative segment decreases and the degeneration of the diseased segment accelerates. Therefore, while decompression of nerve root is completed under total endoscopic nucleus pulposus extraction, tissue engineering of nucleus pulposus is urgently needed to replace the lost part, repair the remaining nucleus pulposus, and enable the disc to be re-sealed and pressurized. Nucleus pulposus tissue engineering is mainly based on cell therapy, and the corresponding biological scaffolds are selected to transplant cells into the diseased area for treatment. However, the current nuclear tissue engineering has some shortcomings, such as limited seed cell source, difficult survival of seed cells, inflammatory rejection in the transplantation area, poor mechanical properties of biological scaffolds, poor degradation performance, and inability to produce biospecific reactions between materials and cells, which seriously restrict the clinical application of nuclear tissue engineering. Human umbilical cord mesenchymal stem cells (hUC-MSCs) are ideal seed cells for the treatment of lumbar disc herniation due to their wide availability, strong proliferation ability and good immune regulation. Therefore, in this project, hUC-MSCs are used for cell transplantation into the vertebral disc of diseased vertebrae. As the treatment method of this project is extremely minimally invasive, it is conducive to the widespread promotion of the technology.

DETAILED DESCRIPTION:
In order to initially observe the safety and effectiveness of human umbilical cord mesenchymal stem cells (hUC-MSCs) transplantation in the treatment of lumbar disc degeneration, this project planned to include a single group of 20 patients with lumbar disc herniation, and adopt an open study design of non-random, self-controlled, single-dose group, and locally inject 2mL hUcMSCs into the lumbar disc of enrolled patients.

The patients were followed up 3, 6 and 12 months after injection to evaluate the safety of hUC-MSCs. Meanwhile, the improvement of patients' low back pain and quality of life were evaluated. Lumbar MRI is used to evaluate the improvement of patients' lumbar disc signal, proving that hUC-MSCs transplantation can delay lumbar disc degeneration and treat lumbar degenerative diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-60 years old;
2. The symptoms are lumbago combined with radiating pain of one lower limb;
3. Failed conservative treatment for 3 months, including physical therapy, manual therapy and non-morphine drug therapy;
4. CT/MRI clearly highlighted the nucleus pulposus pressing the nerve root and the location was consistent;
5. Symptoms and imaging showed unilateral lumbar disc herniation;
6. Imaging showed single-level lumbar disc herniation;
7. MRI (T2WI) of Pfirrmann disc degeneration: Grade I-IV;
8. Lumbar disc herniation segments: L3-4, L4-5, L5-S1;
9. Unilateral full endoscopic extraction of nucleus pulposus;
10. Sign the informed consent;
11. No previous history of spinal surgery.

Exclusion Criteria:

1. Previous history of tumor and spinal infection;
2. Patients with severe coagulation disorders, a history of drug abuse or taking oral anticoagulants;
3. Coma or incapacitation;
4. MRI contraindications (history of cardiovascular and cerebrovascular stent implantation, pacemaker, biostimulator, etc.);
5. Pregnant women;
6. Pregnancy or breastfeeding;
7. Have participated in other clinical trials related to this project within the past 30 days;
8. Those who have received stem cell therapy;
9. Poor compliance, or can not correctly understand the cooperation so that it can not complete the interview;
10. Received intervertebral disc interventional therapy within the past 3 months, such as radiofrequency, laser ablation, protease injection, Ozone injection;
11. Highly allergic or have a history of severe allergies;
12. Patients with severe autoimmune disease or who are receiving immunosuppressive therapy;
13. Serious uncontrolled infection or high fever;
14. Patients with shock, failure of vital organs and unstable vital signs;
15. X-ray showed that the degree of stenosis of the diseased segment was more than 30% compared with the adjacent normal segment;
16. Imaging showed lumbar disc herniation complicated with calcification;
17. Imaging showed lumbar disc herniation with Modic Change;
18. Imaging showed lumbar disc herniation complicated with severe spinal stenosis;
19. Imaging showed lumbar disc herniation complicated with lumbar spondylolisthesis;
20. Imaging showed lumbar disc herniation combined with spinal deformity;
21. Mental disorders, cognitive disorders, or other physical diseases affecting the research results;
22. Doctors believe that there are other reasons for not being included in the treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of lumbar disc MRI (T2WI) signal values | 12 months
  Lumbar MRI images are taken on day 0-1 (measured before stem cell transplantation), 3 months, 6 months and 12 months to record the signal value of the intervertebral disc (4 times in total) from level IV-V to level III and below.

SECONDARY OUTCOMES:
Lower back pain and lower extremity radiating pain relief | 12 months
  VAS scores of low back pain and lower extremity radiative pain are recorded on day 0-1 (measured before stem cell transplantation), 3 months, 6 months, and 12 months (4 times in total) from score 4-10 to score 3 and below.
X-ray Disc Height Index (DHI) | 12 months
  On day 0-1 (measured before stem cell transplantation), 3 months, 6 months, and 12 months, the patients take anterior and lateral lumbar X-rays and record the DHI value (4 times in total) to reach the outcome of DHI≤0.188.
MRI highlights changes in the size of the nucleus pulposus | 12 months
  On day 0-1 (measured before stem cell transplantation), 3 months, 6 months and 12 months, lumbar MRI is taken to measure the size of the protruded nucleus pulposus and record (4 times in total) to reach the outcome of size between 0.7cm×0.5cm×0.5cm and 2.4cm×2.0cm×1.5cm.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No